CLINICAL TRIAL: NCT00281398
Title: Attitudes of Medical Trainees Towards Homeless Persons Presenting for Care in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: 05-31
Record Dates: First submitted 2006-01-18; First posted 2006-01-24 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Homeless Persons; Emergency Medical Services
Keywords: homelessness; Attitudes of medical trainees towards the homeless
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Questionnaire

SUMMARY:
Homelessness is a significant problem in Canada, and many homeless people will seek routine care in the Emergency Department (ED) as a result of barriers to access. There is a paucity of information in the literature concerning the attitudes of health care workers towards homeless patients in the ED setting, although there is ample reason to believe that these attitudes may be suboptimal. In the absence of formal teaching regarding issues of homelessness, medical students have been shown to develop increasingly negative attitudes towards this vulnerable population. It is therefore important to better delineate the attitudes of ED physicians towards homeless persons and to develop an emergency medicine curriculum that helps sensitize physicians to the needs of this already disadvantaged population.

DETAILED DESCRIPTION:
Homelessness increased dramatically in the 1990s and has become a significant problem for Canadian cities. The homeless are at increased risk for both traumatic injuries and serious health problems. Because of significant barriers to access to care, a large proportion of homeless persons will present to the Emergency Department (ED) for acute and routine care. When homeless individuals were asked what was the most difficult aspect of being homeless, negative reactions by shelter workers and health care providers were included as major themes. Despite the recognition that many homeless people are treated in the ED, there is little information regarding the attitudes of ED staff and medical trainees towards these patients and their care. Furthermore, there are no North American curriculum requirements for emergency medicine trainees regarding homelessness or urban health. In the medical setting, exposure alone to homeless patients may negatively impact the attitudes of trainees. We propose to study the attitudes towards homelessness of medical trainees before and after emergency department rotations at an inner city hospital and to define whether implementation of a curriculum on homelessness has a positive impact on attitudes.

This study will be completed over a two year period. During the first year of the study we will survey trainees' attitudes before and after clinical emergency department rotations. We propose to survey the attitudes of medical trainees using the validated questionnaire, the Attitudes Towards Homelessness Inventory (ATHI). A homeless curriculum will be developed using feedback from house staff, health care providers, community partners, and agencies. All undergraduate and postgraduate students will be eligible to participate. In the second year of the study, attitudes will be surveyed before and after completion of the clinical rotation and didactic training.

The primary outcome of interest is to compare the overall ATHI rating of students who are not exposed to the curriculum to those who are exposed. Secondary outcome measures include comparisons of pre and post rotation scores for each trainee. Subgroups will be analyzed according to training program, time of ED rotation, and prior workplace exposure to homeless persons.

ELIGIBILITY:
Inclusion Criteria:

* All undergraduate and postgraduate students will be eligible to participate. In the second year of the study, attitudes will be surveyed before and after completion of the clinical rotation and didactic training.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The main outcome measure is the difference in change in the mean score in those who have participated in the curriculum compared with those who have not during the 2nd year of the study.
Objective 1: To describe the attitudes of medical trainees towards the homeless population before and after completion of an emergency medicine rotation at St. Michael's Hospital
Objective 2: To define, develop, and implement a core curriculum in care of the homeless patient for emergency medicine rotations in Canada
Objective 3: To determine the effect of curriculum implementation on the attitudes of trainees towards homeless patients in the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Julia Spence, MD, FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada